CLINICAL TRIAL: NCT03994796
Title: Genomically-Guided Treatment Trial in Brain Metastases
Brief Title: Genetic Testing in Guiding Treatment for Patients With Brain Metastases
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mirati Therapeutics Inc. (Industry); Genentech, Inc. (Industry); Eli Lilly and Company (Industry); Kazia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A071701; NCI-2019-00744 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2019-06-14; First posted 2019-06-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: CDK Gene Mutation; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm; NTRK Family Gene Mutation; PI3K Gene Mutation; ROS1 Gene Mutation; KRAS G12C Mutation
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; entrectinib; adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (CDK gene mutation) (Experimental): Patients receive abemaciclib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib
- Arm II (PI3K gene mutation) (Experimental): Patients receive PI3K inhibitor paxalisib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PI3K Inhibitor paxalisib
- Arm III (NTRK/ROS1 gene mutation) (Experimental): Patients receive entrectinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Entrectinib
- Arm IV (KRAS G12C mutation) (Experimental): Patients receive adagrasib (MRTX849) PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adagrasib

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Arms: Arm I (CDK gene mutation)
Drug: PI3K Inhibitor paxalisib — Given PO
  Arms: Arm II (PI3K gene mutation)
Drug: Entrectinib — Given PO
  Arms: Arm III (NTRK/ROS1 gene mutation)
Drug: Adagrasib — Given PO
  Other Names: MRTX849
  Arms: Arm IV (KRAS G12C mutation)

SUMMARY:
This phase II trial studies how well genetic testing works in guiding treatment for patients with solid tumors that have spread to the brain. Several genes have been found to be altered or mutated in brain metastases such as NTRK, ROS1, CDK, PI3K, or KRAS G12C. Medications that target these genes such as abemaciclib, paxalisib, entrectinib and adagrasib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Genetic testing may help doctors tailor treatment for each mutation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the activity of a CDK inhibitor in patients with progressive brain metastases derived from lung cancer, breast cancer, and other cancers harboring actionable genetic alterations associated with sensitivity to CDK inhibitors as measured by response rate (Response Assessment in Neuro-Oncology [RANO] criteria).

II. To determine the activity of a PI3K inhibitor in patients with progressive brain metastases derived from lung cancer, breast cancer, and other cancers harboring actionable genetic alterations in the PI3K pathway as measured by response rate (RANO criteria).

III: To determine the activity of an NTRK/ROS1 inhibitor in patients with progressive brain metastases derived from lung cancer harboring actionable NTRK/ROS1 gene fusions as measured by response rate (RANO criteria).

IV. To determine the activity of an KRAS G12C inhibitor in patients with progressive brain metastases derived from lung cancer, and other cancers harboring a KRAS G12C mutation as measured by response rate (RANO criteria).

SECONDARY OBJECTIVES:

I. To evaluate the systemic response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria in each of the cohorts determined by treatment and primary cancer type.

II. To evaluate the clinical benefit rate (complete response [CR] + partial response [PR] + stable disease [SD]) by Brain Metastases (BM)-RANO for central nervous system (CNS) in each of the cohorts determined by treatment and primary cancer type.

III. To evaluate the clinical benefit rate (CR + PR + SD) by RECIST for extracranial disease in each of the cohorts determined by treatment and primary cancer type.

IV. To evaluate the duration of response by BM-RANO in each of the cohorts determined by treatment and primary cancer type.

V. To evaluate the duration of response by RECIST in each of the cohorts determined by treatment and primary cancer type.

VI. To evaluate the progression-free survival for intracranial disease in each of the cohorts determined by treatment and primary cancer type.

VII. To evaluate the progression-free survival for extracranial disease in each of the cohorts determined by treatment and primary cancer type.

VIII. To evaluate the site of first progression (CNS versus [vs] non-CNS) in each of the cohorts determined by treatment and primary cancer type.

IX. To evaluate the overall survival in each of the cohorts determined by treatment and primary cancer type.

X. To evaluate the toxicity profile of agents in patients with brain metastases in each of the cohorts determined by treatment and primary cancer type.

OUTLINE: Patients are assigned to 1 of 4 arms.

ARM I (CDK GENE MUTATION): Patients receive abemaciclib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II (PI3K GENE MUTATION): Patients receive PI3K inhibitor paxalisib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM III (NTRK/ROS1 GENE MUTATION): Patients receive entrectinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM IV (KRAS G12C MUTATION): Patients receive adagrasib (MRTX849) PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 8 weeks for 2 years, then every 3 months for years 3-4, and then every 6 months thereafter for up to 5 years after registration.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION ELIGIBILITY CRITERIA (ALL PATIENTS) • Tissue available for biomarker testing (any brain metastasis tissue and extracranial site from any prior resection or biopsy).

REGISTRATION ELIGIBILITY CRITERIA (ALL PATIENTS)

* Participants must have histologically confirmed parenchymal metastatic disease to the brain from any solid tumor. Note: this includes patients that have controlled extracranial disease with progressive intracranial metastasis, as well as patients that have progressive intracranial and extracranial disease.
* New or progressive brain metastases are defined as any one of the following:

  * Untreated measurable lesions in patients who have received surgery and/or stereotactic radiosurgery (SRS) to one or more other lesions.
  * Progressive measurable lesions after radiation, surgery, or prior systemic therapy
  * Residual or progressive lesions after surgery if asymptomatic.
  * Patients who have had prior whole-brain radiotherapy (WBRT) and/or SRS and then whose lesions have progressed by BM-RANO criteria or there are new lesions, are eligible. Lesions treated with SRS may be eligible if there is unequivocal evidence of progression. For patients with NTRK or ROS1 mutations, entrectinib may be used for newly diagnosed brain metastases. Similarly, for patients with KRAS G12C mutations, MRTX849 may be used for newly diagnosed brain metastases.
  * Patients who have not previously been treated with cranial radiation (e.g. WBRT or SRS) are eligible, but such patients must be asymptomatic or neurologically stable from their CNS metastases.
* Measurable CNS disease (=> 10 mm).
* Ability to obtain magnetic resonance imaging (MRI)s with contrast
* No surgery within 2 weeks prior to or after registration.
* No chemotherapy within 14 days prior to registration (Note: for abemaciclib arm, a 21-day chemotherapy washout is required).

  * For melanoma, patients must have progressed after prior immune checkpoint blockade or for BRAF positive melanoma, BRAF/MEK inhibitors.
  * For lung cancer, EGFR mutant patients must have failed EGFR therapies
  * For HER2-positive breast cancer patients (regardless of ER/PR status), patients must have received at least one prior HER-2 directed therapy in the metastatic setting.
  * For triple negative breast cancer (TNBC), patients must have received at least one chemotherapy in the metastatic setting.
  * For estrogen receptor (ER) and/or progesterone receptor (PR)+ HER2-negative breast cancer, patients must have received at least one endocrine therapy in the metastatic setting.
  * Patients who have received prior treatment with any of the targeted treatments on this study are not eligible for that specific treatment arm(s), but could be eligible for other arms (e.g., a patient who has had prior treatment with abemaciclib would not be eligible for the abemaciclib arm, but could be eligible for another arm).
* Presence of clinically actionable alteration in NTRK, ROS1, KRAS G12C or CDK pathway or PI3K pathway in both a brain metastasis and extracranial site per central review.
* Not pregnant and not nursing, because this study involves investigational agents whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required (Note: for abemaciclib arm, pregnancy test is required =< 7 days prior to registration).
* No known current diffuse leptomeningeal involvement for the CDK, PI3K and NTRK arms (diffuse defined as leptomeningeal involvement throughout the CNS axis).Patients with focal leptomeningeal disease, with or without documented positive CSF cytology, are eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate organ function.
* Absolute neutrophil count (ANC) >= 1,500/mm^3.
* Platelet count >= 100,000/mm^3.
* Total bilirubin =< 1.5 x upper limit of normal (ULN) except in patients with Gilbert's disease. Patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN).
* Creatinine =< 1.5 mg/dL OR calculated (Calc.) creatinine clearance > 45 mL/min except for patients in the adagrasib (MRTX849) (KRAS G12C) arm. For this arm, patients must have creatinine clearance ≥60 mL/min or glomerular filtration rate ≥60 mL/min/1.73m2 calculated using a validated prediction equation (e.g., Cockcroft-Gault, MDRD, or 24-hour urine CrCl).
* No uncontrolled medical comorbidities per investigator discretion (e.g. interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea)
* Radiation to symptomatic non-target sites within neural axis is allowed prior to registration without washout (provided there is at least one untreated target lesion for measurement on study and radiation is completed prior to registration).
* Concurrent systemic corticosteroids are allowed if stable dose of dexamethasone for 7 days prior to registration. Baseline doses and changes in steroid dosing will be captured.
* No concurrent administration of anticancer therapies (except for endocrine therapy or continuation of hormonal therapy or trastuzumab in breast cancer patients for the PI3K and CDK inhibitor arms). . No chemotherapy, targeted therapy or immunotherapy within 14 days prior to entering the study (Note: For abemaciclib arm, a 21-day chemotherapy washout is required).
* Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug 14 days or 5 or more half-lives prior to registration on the study.
* Chronic concomitant treatment with strong CYP3A4 inducers is not allowed. Patients must discontinue the drug 14 days prior to the start of study treatment.

ADDITIONAL REGISTRATION ELIGIBILITY CRITERIA FOR PAXALISIB ARM

* Urine protein to creatinine (UPC) ratio < 1 or urine protein =< 1.
* Recent acute myocardial infarction in the last 6 months or current angina pectoris are excluded. Patients with symptomatic bradycardia should have an electrocardiogram at baseline. If QT interval > 470 msec, the patient is excluded.
* Patients with uncontrolled type I or II diabetes mellitus should be excluded. Uncontrolled diabetes is defined as glycosylated hemoglobin (HbA1c) > 9% in addition to fasting glucose > 140 mg/dL on at least 2 occasions within 14 days prior to registration.

ADDITIONAL REGISTRATION ELIGIBILITY CRITERION FOR ENTRECTINIB ARM

• Concurrent use of H2 receptor antagonists, receptor antagonists, proton pump inhibitors (PPIs), and/or antacids are prohibited.

ADDITIONAL REGISTRATION ELIGIBILITY CRITERION FOR ABEMACICLIB ARM

* Hemoglobin >= g/dL. Patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
* Patients who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to registration. A washout period of at least 21 days is required between last chemotherapy dose and registration (provided the patient did not receive radiotherapy).
* Patients who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and registration.
* Breast cancer patients who have received ribociclib or palbociclib are eligible as long as there is documentation of CDK4/6 pathway alteration on a biopsy or resection at the point of progression post-ribociclib or palbociclib.
* For females of childbearing potential: A female of childbearing potential, must have a negative serum pregnancy test within 7 days prior to registration and agree to use a highly effective contraception method during the treatment period and for 3 weeks following the last dose of abemaciclib. Contraceptive methods may include an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection. Cases of pregnancy that occur during maternal exposures to abemaciclib should be reported. If a patient or spouse/partner is determined to be pregnant following abemaciclib initiation, she must discontinue treatment immediately. Data on fetal outcome and breast-feeding are to be collected for regulatory reporting and drug safety evaluation.
* Patients with active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive] are excluded. Screening is not required for enrollment.
* Patients with personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest, are excluded.

ADDITIONAL REGISTRATION ELIGIBILITY CRITERION FOR ADAGRASIB (MRTX849) ARM

* Hemoglobin ≥9.0 g/dL. Note: Transfusions will be allowed to achieve this provided the patient has not received more than 2 units of red blood cells in the prior 4 weeks.
* Any of the following cardiovascular abnormalities within 6 months of study entry are excluded: symptomatic or uncontrolled atrial fibrillation, unstable angina pectoris or myocardial infarction, CHF ≥ NYHA Class 3, stroke or transient ischemic attack.
* Ongoing need for medication known to cause prolonged QTc interval or that are substrates of CYP3A4 with narrow therapeutic index that cannot be switched to alternative treatment prior to study entry is excluded.
* Prolonged QTc interval >480 milliseconds or family history or medical history of Long QT syndrome is excluded.•
* Known human immunodeficiency virus (HIV) infection or acute or chronic hepatitis B or C infection is excluded. Screening is not required for enrollment. Note that the following are permitted:

  * Patients treated for hepatitis C (HCV) with no detectable viral load;
  * Patients treated for HIV with no detectable viral load for at least 1 month prior to randomization while on a stable regimen of agents that are not strong inhibitors of CYP3A4; and
  * Patients with hepatitis B (HBV) receiving prophylaxis against reactivation of hepatitis B (either [HBsAg-positive with normal ALT and HBV DNA <2,000 IU/mL or <10,000 copies/mL] or [HBsAg-negative and anti-HBc positive]).
* History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow oral medications is excluded.
* Recovery from the adverse effects of prior therapy to baseline or Grade 1 (any grade alopecia and Grade ≤2 peripheral neuropathy are eligible).
* For females of childbearing potential. It is not known whether MRTX849 presents a risk to the embryo or the fetus; however, based on the mechanism of action (KRAS G12C inhibition), effects on the reproductive system are not unexpected. MRTX849 is contraindicated in women who are pregnant or lactating. Women of childbearing potential and men receiving MRTX849 who are sexually active must employ an effective method of contraception throughout their period of treatment and for 6 months after their last treatment with MRTX849.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate in the brain | Up to 5 years
  Assessed per Response Assessment in Neuro-Oncology (RANO) criteria for brain metastases. The response rate is defined as the number of patients who have achieved complete response (CR) or partial response (PR) per RANO for brain metastases criteria during treatment with CDK, PI3K, NTRK/ROS, or KRAS G12C inhibitors divided by total number of evaluable patients. The response rate and associated exact confidence interval will be estimated within each cohort defined by the targeted agent and histology.

SECONDARY OUTCOMES:
Systemic response for extracranial disease | Up to 5 years
  Assessed with Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Will be estimated using the systemic response rate (SRR) - where SRR is defined as the number of evaluable patients achieving a response (PR or CR per RECIST 1.1) during treatment with study therapy divided by the total number of evaluable patients. Point estimates will be generated for systemic response rates within each cohort with corresponding 95% binomial confidence intervals.
Clinical benefit rate for central nervous system (CNS) | Up to 5 years
  Evaluated by Response Assessment in Neuro-Oncology (RANO) criteria. Will be estimated as the number of evaluable patients achieving stable disease (SD), partial response (PR), or complete response (CR) as their best objective response during treatment with protocol therapy divided by the total number of evaluable patients. Point estimates will be generated for clinical benefit rates within each cohort with corresponding 95% binomial confidence intervals.
Clinical benefit rate for extracranial disease | Up to 5 years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST). Will be estimated as the number of evaluable patients achieving stable disease (SD), partial response (PR), or complete response (CR) as their best objective response (per RECIST for extracranial disease) during treatment with protocol therapy divided by the total number of evaluable patients. Point estimates will be generated for clinical benefit rates within each cohort with corresponding 95% binomial confidence intervals.
Duration of response for brain metastases | From the time measurement criteria are met for CR or PR for brain metastases until the first date that progressive CNS disease or death is documented, assessed up to 5 years
  Duration of response for brain metastases is defined for all evaluable patients who have achieved a confirmed response as the time from the date at which the patient's objective status for brain metastases is first noted to be a CR or PR (per Response Assessment in Neuro-Oncology [RANO] for brain metastases) to the date of the earliest progressive CNS disease is documented or death. The median and 95% confidence intervals will be estimated using the Kaplan-Meier estimator. No formal comparison will be made among the cohorts.
Duration of response for extracranial disease | From the time measurement criteria are met for CR or PR for extracranial disease until the first date that progressive disease for extracranial disease or death is documented, assessed up to 5 years
  Duration of response for extracranial disease is defined for all evaluable patients who have achieved a confirmed response as the time from the date at which the patient's objective status for extranial disease is first noted to be a CR or PR (per RECIST1.1) to the date of the earliest progression (PD) for extracranial disease is documented or death. The median and 95% confidence intervals will be estimated using the Kaplan-Meier estimator. No formal comparison will be made among the cohorts.
Progression-free survival (PFS) - intracranial | From first day of study treatment to the earliest date documentation of intracranial disease progression or death from any cause, assessed up to 5 years
  Intracranial PFS is defined as the time from the first day of study treatment to the earliest date of intracranial disease progression (per RANO for brain metastases) or death from any cause, whichever comes first. The median and 95% confidence intervals will be estimated using the Kaplan-Meier estimator. No formal comparison will be made among the cohorts.
Progression-free survival (PFS) - extracranial | From the first day of study treatment to the earliest date of documentation of extracranial disease progression or death from any cause, assessed up to 5 years
  Extracranial PFS is defined as the time from the first day of study treatment to the earliest date of extracranial disease progression (per RECIST1.1) or death from any cause, whichever comes first. The median and 95% confidence intervals will be estimated using the Kaplan-Meier estimator. No formal comparison will be made among the cohorts.
Site of first progression | Up to 24 months
  The site of first progression will be estimated descriptively within each cohort within 12 and 24 months after starting protocol treatment. The first progression is defined as the first documented central nervous system (CNS) progression per Response Assessment in Neuro-Oncology (RANO) or extracranial progression per Response Evaluation Criteria in Solid Tumors (RECIST), whichever occurs first. The percentage of extracranial progression at first progression within 12 and 24 months after starting protocol treatment will be estimated as number of patients who experience the first progression which is extracranial progression divided by number of patients who are still at risk up to 12 and 24 months, respectively.
Overall survival | From the first day of study treatment to death due to any cause, assessed up to 5 years
  Overall survival is defined as the time from the first day of study treatment to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. No formal comparison will be made among the cohorts.
Incidence of adverse events | Up to 5 years
  Assessed per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, toxicity is defined as adverse events that are classified as possibly, probably, or definitely related to study treatment. Toxicities will be evaluated via the ordinal CTCAE standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by patient and treatment cohort will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of the analysis. No formal comparison will be made among the cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Brastianos, MD, Study Chair — Massachusetts General Hospital
Locations (435):
- United States (435):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner LSU Health Saint Mary's Medical Center, Shreveport, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Memorial Hermann Northeast Hospital, Humble, Texas
  - Memorial Hermann The Woodlands Hospital, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sammons S, Van Swearingen AED, Anders CK. Receptor discordance in breast cancer brain metastases: when knowledge is power. Neuro Oncol. 2020 Aug 17;22(8):1060-1061. doi: 10.1093/neuonc/noaa131. No abstract available. PMID 32479604